CLINICAL TRIAL: NCT00116662
Title: A Single-Blind, Dose-Escalating Study to Assess Efficacy and Safety of Resiquimod Gel Applied 3 Times Per Week for up to 12 Weeks for the Treatment of Common Warts in Pediatric Subjects
Brief Title: An up to Twelve Week Safety and Efficacy Study With a Topical Gel to Treat Common Warts in Pediatric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1534-RESI
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2006-11

CONDITIONS: Warts
Keywords: Wart(s); Common Wart(s); Children; Pediatric; 3M Pharmaceuticals; Resiquimod
MeSH Terms: conditions — Warts | interventions — resiquimod

INTERVENTIONS:
Drug: Resiquimod

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness in pediatric subjects of three different strengths of resiquimod gel applied to common wart(s) three times a week for up to twelve weeks.

A second purpose is to evaluate the safety of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of common wart(s)
* Ages between 3 to 11

Exclusion Criteria:

* Other types of wart(s), ie. plantar
* Currently participating in another clinical study
* Chronic viral hepatitis B or C

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84
Dates: Start 2005-03

PRIMARY OUTCOMES:
Clearance of treated common wart(s)

SECONDARY OUTCOMES:
Partial clearance of treated common wart(s)
Wart recurrence

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Arkansas, Fayetteville, Arkansas
  - Arkansas, Little Rock, Arkansas
  - Georgia, Newnan, Georgia
  - Illinois, Buffalo Grove, Illinois
  - Indiana, Lafayette, Indiana
  - Kansas, Wichita, Kansas
  - Massachusetts, Boston, Massachusetts
  - Missouri, St Louis, Missouri
  - Utah, Layton, Utah
  - Vermont, Burlington, Vermont